CLINICAL TRIAL: NCT04860440
Title: A Feasibility Study of a Wrist Worn Accelerometer to Characterise the Physical Activity of Patients With End-stage Renal Disease (W-WARD Study).
Brief Title: A Study of Wrist Worn Accelerometers in End-Stage Renal Disease
Acronym: W-WARD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, James Richards, Academic Clinical Lecturer & Senior Clinical Fellow in HPB & Transplantation Surgery, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: W-WARD2020v1
Record Dates: First submitted 2021-04-14; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Chronic Kidney Diseases; End Stage Renal Disease on Dialysis; Frailty
MeSH Terms: conditions — Renal Insufficiency, Chronic; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- End-Stage Renal Disease on haemodialysis: Wearing accelerometer (fitness tracker) for 7 days.
  Interventions: Device: GeneActiv wrist worn accelerometer
- Low clearance pre-dialysis patients: Wearing accelerometer (fitness tracker) for 7 days.
  Interventions: Device: GeneActiv wrist worn accelerometer

INTERVENTIONS:
Device: GeneActiv wrist worn accelerometer — Wrist worn device worn for 7 days

SUMMARY:
The kidneys are important at getting rid of toxins and excess water from the body. If they fail, then toxins and excess water builds up within the body. Kidney failure is treated by either giving patients a new kidney (a transplant) or by removing the toxins and fluid from the body by the process of dialysis.

The investigators' aim is to personalise the care given to patients with kidney failure, and as such, they have started measuring the fitness of patients with kidney failure, who either already require dialysis or may need dialysis in the near future. This is currently done in a number of ways including measuring how strong their grip is, assessing their walking speed and asking questions about how difficult they find certain activities.

In the future, the investigators think that this will allow targeted treatments to help improve their fitness and potentially identify any problems earlier.

Current approaches to measuring activity and fitness have limitations and in particular may over- or underestimate the level of the physical activity. To over come these limitations, participants will be asked to wear an activity tracker (called an accelerometer) on for a week. Readings from the accelerometer will be compared against the other markers of fitness and activity to see if they are comparable. It will also be noted whether patients are prepared to wear the device for 7 days (compliance).

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18 years with low clearance pre-dialysis and referred to the Low Clearance Clinic with estimated Glomerular Filtration Rate (eGFR) less than 20 ml/min/1.73m and / or commenced on haemodialysis
2. Able to give informed consent

Exclusion Criteria:

1. Significant resting tremor of any aetiology or severe Parkinson's Disease
2. Immobile
3. Arteriovenous fistulas in both arms
4. Any scheduled inpatient treatment or day case treatment in next 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Low clearance pre-dialysis patients referred to the Low Clearance Clinic and / or who have commenced on haemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 7 days
  The acceptability of physical activity measures in frailty assessment in patients from the low clearance and dialysis clinic as determined by the percentage of time, device worn during the 7-day period.

SECONDARY OUTCOMES:
Measurement of physical activity by the accelerometer | 7 days
  Measurement of physical activity by the accelerometer (no units)
Fried Frailty Phenotype (no units) | 1 day
  Fried Frailty Phenotype (no units)
Grip strength (in kilograms) | 1 day
  Grip strength (in kilograms)
Walking speed (in seconds measured over 15 feet) | 1 day
  Walking speed (in seconds measured over 15 feet)
Clinical Frailty Scale (no units) | 1 day
  Clinical Frailty Scale (no units)
10 Point Cognitive Screener (no units) | 1 day
  10 Point Cognitive Screener (no units)
4AT Assessment Tool of Cognitive Impairment (no units) | 1 day
  4AT Assessment Tool of Cognitive Impairment (no units)

CONTACTS AND LOCATIONS:
Overall Officials: James A Richards, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- James Richards, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No